CLINICAL TRIAL: NCT03485326
Title: A Multi-Centre, Prospective, Non-Interventional Study to Intensively Monitor the Safety of Osimertinib in Clinical Practice Among Chinese NSCLC Patients An Observational Study Conducted Among Chinese NSCLC Patients to Evaluate Osimertinib Safety Profile in a Real World Setting
Brief Title: A Multi-Centre, Prospective, Non-Interventional Study to Intensively Monitor the Safety of Osimertinib in Clinical Practice Among Chinese NSCLC Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00026
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Osimertinib; Tagrisso; NSCLC; Non-small cell lung cancer; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Safety: Safety

SUMMARY:
This is a multi-center, prospective, non-interventional study. The study will enroll about 1700 Chinese patients diagnosed as NSCLC and treated with osimertinib at least one dose.

The objective of this non-interventional study is to monitor the safety profile of osimertinib in Chinese NSCLC patients in real world clinical practice.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-interventional study. The study will enroll about 1700 Chinese patients diagnosed as NSCLC and treated with osimertinib at least one dose. The investigator in an observational study cannot intervene in the treatment. The prescribing doctor is in charge of prescribing or discontinuation of osimertinib. It is planned that all eligible patients who received at least one dose of osimertinib at the participating sites will be enrolled until 1700 patients has been recruited.

The recruited patients will be followed up according to standard clinical practice. They will be tracked up to 30 days after discontinuation of osimertinib treatment, or 12 months after study enrolment, whichever comes earlier. For patients who accrued SAE, the SAE will be followed up until the outcome is defined, or the study is terminated, whichever comes earlier. The study would be terminated 12 months after the last patient is enrolled.

The objective of this non-interventional study is to monitor the safety profile of osimertinib in Chinese NSCLC patients in real world clinical practice.

The primary endpoint of this study is the incidence of all adverse drug reactions (ADRs). The second endpoints include the severity for AEs, the incidence of all AEs, AESIs, SAEs, the incidence of AEs for elderly population (age ≥ 65 years old), and AEs leading to osimertinib-associated interruption, dose reduction, discontinuation, and death

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
* Patients histologically or cytologically diagnosed as NSCLC
* Eligible for osimertinib treatment per the judgement of the treating physician in clinical practice
* Received at least one dose of osimertinib

Exclusion Criteria:

• Enrollment in other on-going studies, which prohibit any participation in this non-interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit about 1700 Chinese patients histologically or cytologically diagnosed as NSCLC and received at least one dose of osimertinib treatment in China mainland.
Sampling Method: Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Incidence of all ADRs | From time of patients enrolled in the study until end of study follow-up (30 days after discontinuation of osimertinib treatment, or 12 months after study enrolment, whichever comes earlier)
  Incidence of all Adverse drug reaction

CONTACTS AND LOCATIONS:
Overall Officials: Baohui HAN, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (21):
- China (21):
  - Research Site, Beijing
  - Research Site, Chengde
  - Research Site, Chengdu
  - Research Site, Dingzhou
  - Research Site, Fuzhou
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Huanghua
  - Research Site, Jinan
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Weihai
  - Research Site, Wuhan
  - Research Site, Zhuji

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zhong H, Jiang S, Yao W, Song X, Lv D, Zhu D, Guo Y, Ding C, Xue Y, Bai X, Xiao L, Chen P, Wang Y, Tian P, Lin G, Li W, Chen J, Hu Y, Xia B, Wang Z, Long H, Yao W, Zhang H, Zhao Q, Wang Y, Lu L, Duan W, Xing L, Yang F, Chen Y, Wei Y, Han B, He J. Safety of osimertinib in Chinese patients with non-small cell lung cancer: a multi-center, prospective, observational study. Future Oncol. 2025 Dec;21(28):3639-3648. doi: 10.1080/14796694.2025.2579208. Epub 2025 Oct 30. PMID 41164890
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00026&attachmentIdentifier=5665c5e9-0f9d-445d-b1a6-a02cb0b130ad&fileName=Tagrisso_DIM-CSR_Synopsis_redact.pdf&versionIdentifier=